CLINICAL TRIAL: NCT01160562
Title: Pilot Study to Estimate the Burden and Distribution of Plasmodium Falciparum Malaria in Kalifabougou, Mali in Preparation for a Prospective Cohort Study of Naturally-Acquired Malaria Immunity
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910155; 10-I-N155
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-01-23

CONDITIONS: Malaria, Falciparum; Plasmodium Falciparum
Keywords: Prevalence; Incidence; Children; Adults; Global Positioning system
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Plasmodium falciparum malaria remains a global public health threat. Leading malaria vaccine candidates confer only partial short-lived protection at best. An understanding of the mechanisms by which humans acquire malaria immunity through repeated P. falciparum infections may aid the development of a malaria vaccine. This pilor study is designed to initiate the epidemiological groundwork for a future prospective cohort study of acquired malaria immunity in Kalifabougou, Mali, a rural village of approximately 5 000 individuals who are exposed to seasonal P. falciparum transmission each year from July through December. This study will estimate the age-stratified point prevalence of P. falciparum infection before the malaria season and at the peak of the 6-month malaria season, and it will estimate the age-stratified incidence of symptomatic p. falciparum infection during the 6-month malaria season. The spatial distribution of asymptomatic P. falciparum infections and incident malaria cases within the village of Kalifabougou will be determined by merging the prevalence and incidence data with census and Global Positioning System (GPS) data....

DETAILED DESCRIPTION:
Plasmodium falciparum malaria remains a global public health threat. Leading malaria vaccine candidates confer only partial short-lived protection at best. An understanding of the mechanisms by which humans acquire malaria immunity through repeated P. falciparum infections may aid the development of a malaria vaccine. This pilor study is designed to initiate the epidemiological groundwork for a future prospective cohort study of acquired malaria immunity in Kalifabougou, Mali, a rural village of approximately 5 000 individuals who are exposed to seasonal P. falciparum transmission each year from July through December. This study will estimate the age-stratified point prevalence of P. falciparum infection before the malaria season and at the peak of the 6-month malaria season, and it will estimate the age-stratified incidence of symptomatic p. falciparum infection during the 6-month malaria season. The spatial distribution of asymptomatic P. falciparum infections and incident malaria cases within the village of Kalifabougou will be determined by merging the prevalence and incidence data with census and Global Positioning System (GPS) data.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cross-sectional Survey:

Individuals (ages 2-25 years) are eligible to enter the cross-sectional study if they agree to:

* Live in Kalifabougou for the next 5 months.
* Have blood specimens stored for future studies.

Passive Surveillance:

All individuals who live in Kalifabougou and present to the Kalifabougou health center with suspected malaria will be eligible to enroll in the passive surveillance component of the protocol.

EXCLUSION CRITERIA:

None.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1719 (Actual)
Dates: Start 2010-06-23; Study Completion 2013-01-23

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Crompton, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Vekemans J, Ballou WR. Plasmodium falciparum malaria vaccines in development. Expert Rev Vaccines. 2008 Mar;7(2):223-40. doi: 10.1586/14760584.7.2.223. PMID 18324891
- [Background] Langhorne J, Ndungu FM, Sponaas AM, Marsh K. Immunity to malaria: more questions than answers. Nat Immunol. 2008 Jul;9(7):725-32. doi: 10.1038/ni.f.205. PMID 18563083
- [Background] Crompton PD, Traore B, Kayentao K, Doumbo S, Ongoiba A, Diakite SA, Krause MA, Doumtabe D, Kone Y, Weiss G, Huang CY, Doumbia S, Guindo A, Fairhurst RM, Miller LH, Pierce SK, Doumbo OK. Sickle cell trait is associated with a delayed onset of malaria: implications for time-to-event analysis in clinical studies of malaria. J Infect Dis. 2008 Nov 1;198(9):1265-75. doi: 10.1086/592224. PMID 18752444